CLINICAL TRIAL: NCT06543199
Title: Evaluation of the Effect of Hypericum Perforatum L and Hyaluronic Acid on Excisional
Brief Title: Evaluation of the Effect of Hypericum Perforatum L and Hyaluronic Acid on Excisional Palatal Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Tugba Aydin, associate professor doctor, Ataturk University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 421
Record Dates: First submitted 2024-08-04; First posted 2024-08-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Wound Healing Disorder; Palate; Wound
Keywords: palatal wound healing; hyaluronic acid; Hypericum perforatum L
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CONTROL (Experimental): Group in which no agent was used in the area left for secondary healing at the donor site.
  Interventions: Procedure: wound healing monitoring
- HYPERICUM PERFORATUM L (Experimental): Group using hypericum perforatum L agent in the area left for secondary healing at the donor site.
  Interventions: Procedure: Local application of hypericum perforatum L to the wound site; Procedure: wound healing monitoring
- HYALURONIC ASID (Experimental): Group using hyaluronıc acid agent in the area left for secondary healing at the donor site.
  Interventions: Procedure: local application of hyaluronic acid agent to the wound site; Procedure: wound healing monitoring

INTERVENTIONS:
Procedure: local application of hyaluronic acid agent to the wound site — Evaluation of the effect of local use of hyaluronic acid agent on wound healing
  Arms: HYALURONIC ASID
Procedure: Local application of hypericum perforatum L to the wound site — Hyperıcum perforatum L ajanının lokal kullanımının yara iyileşmesine etkisinin değerlendirilmesi
  Arms: HYPERICUM PERFORATUM L
Procedure: wound healing monitoring — Doctor visit on days 3, 7, 14, 21 and 28

SUMMARY:
The free gingival graft (FGG) procedure is one of the surgical approaches used to create a large area of adherent gingiva around the tooth and implant. As part of this procedure, one SDG at a time is harvested from the donor site of the secondary healing palate. The most common postoperative complications are pain, burning sensation and delayed wound healing at the donor site. Many agents have been used for years to reduce these complications, but so far none has been emphasized as the ideal agent. In this thesis, methods to improve the healing of the hard palate, the donor site for SDG surgery, and postoperative patient comfort will be compared.

DETAILED DESCRIPTION:
The free gingival graft (FGG) procedure is one of the surgical approaches used to create a large adherent gingival and keratinized zone around teeth and implants. As part of this procedure, SDG is harvested from the palatal donor area. The most common postoperative complications from the palatal donor area left to secondary healing are pain, burning sensation and delayed wound healing at the donor site. Various hemostatic agents, dressing materials, platelet-rich fibrin and analgesics have been used for years to reduce postoperative complications, promote wound healing and increase patient comfort. However, none of them has been emphasized as the ideal agent in the relevant literature. In this thesis, we will compare the methods that will improve the healing of the hard palate, which is the donor site for SDG surgery, and postoperative patient comfort. Hypericum perforatum L and hyaluronic acid will be compared by local application to the palatal rotator area.

It is aimed to investigate the postoperative effects of topical application of Hypericum perforatum L and hyaluronic acid (trade names; HYPERICUM PERFORATUM L Dr Özberk St. John's wort oil; hyaluronic acid: Gengigel Forte Gel) on the healing of surgical wounds created in the palatal donor area after SDG and its effects on wound healing. Hyaluronic acid is a non-sulfated polysaccharide component of the glycosaminoglycan family, which is also found in joint fluids, serum and various body fluids such as saliva and gingival groove fluid. Although it is present in all periodontal tissues, it is especially prominent in non-mineralized tissues such as gingiva and periodontal ligament. The highly biocompatible and nonimmunogenic nature of the action of hyaluronic acid, its bacteriostatic, fungistatic, anti-inflammatory, antiedematous, osteoinductive and pro-angiogenetic properties leading to the promotion of wound healing in various tissues have led hyaluronic acid to be of interest in the treatment of various diseases in medical fields such as orthopedics, ophthalmology and dermatology. In dentistry, hyaluronic acid has been used in tooth extraction sockets, temporomandibular joint treatment to accelerate the healing process and to make the healing period comfortable.

Plants have always played an important role in the improvement of human health in history. Hypericum perforatum, a member of the Hypericaceae family, has been recognized as a valuable herbal medicine. This plant contains hyperforin, flavonoids and hypericin. The olive oil extract of H. perforatum has long been used as both topical and oral medicine to treat cuts, burns, depression, hemorrhoids, diabetes and gastrointestinal ulcers. Studies have shown that H. perforatum increases collagen deposition, shortens the duration of inflammation and stops the migration of fibroblasts during wound healing.

Both agents have many areas of use that have been tried and found to be effective on wound healing. It is aimed to contribute to the literature by evaluating these two agents in terms of wound healing and postoperative patient comfort in the palatal donor area and at the same time evaluating them with a control group in which no agent was used.

ELIGIBILITY:
Inclusion Criteria:

* The patient is in need of free gingival graft (FGG) surgery,
* The patient's acceptance of the treatment,
* All oral plaque and bleeding scores less than 20%.
* Age between 18-60 years.

Exclusion Criteria:

* The patient does not need SDG surgery,
* The patient is a smoker,
* The patient has a systemic disease that will affect recovery,
* The patient is unable to attend follow-up sessions,
* Previous periodontal surgery,
* The patient is pregnant or lactating,
* The patient has used antibiotics, corticosteroids, anti-inflammatory, immunosuppressive drugs in the last 6 months.
* Tooth deficiency such that the patient cannot wear acrylic aligners
* Acute periodontal condition

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — the fact that wound healing in the oral region is more difficult in women compared to men in this surgery.
Enrollment: 45 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
assessment of pain at the donor site | Days 1,2,3,4,4,5,6,7
  Measuring and recording the pain score at the donor site with a vas
evaluation of burning in the donor area | Days 1,2,3,4,4,5,6,7
  Measuring and recording the burning score at the donor site with a vas
evaluation of chewing discomfort at the donor site | Days 1,2,3,4,4,5,6,7
  Measuring and recording the chewing discomfort score at the donor site with a vas

CONTACTS AND LOCATIONS:
Locations (1):
- Tuğba Aydın, Erzurum, Hiçbiri Seçilmedi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes